CLINICAL TRIAL: NCT05261373
Title: Efficacy of a Nutritional Education Strategy and Role of Physical Exercise on the Modulation of Muscle Metabolism Through the Gut Microbiota in Type 2 Diabetics (THE EDUGUTION PROJECT)
Brief Title: Efficacy of a Nutritional Education Strategy and Physical Exercise on the Gut Microbiota in Type 2 Diabetics
Acronym: EDUGUTION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cadiz (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The EDUGUTION project
Record Dates: First submitted 2021-12-17; First posted 2022-03-02 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases; Fat Burn; Metabolism Disorder
Keywords: Gut microbiota; High intensity interval training; Insulin resistance; Diet; Fat metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Metabolic Diseases; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: The project is a randomized controlled clinical trial with T2DM and obesity
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control (CG+INACT) (No Intervention): Participants who do not receive neither nutritional education nor exercise program. They will be instructed to maintain their normal life habits with respect to physical activity and diet.
- Moderate-intensity continuous training (CG+MICT) (Active Comparator): Participants who do not receive nutritional education but are enrolled in a moderate-intensity continuous training exercise program.
  Interventions: Other: The Moderate-Intensity Continuous Training (MICT)
- High-intensity interval training (CG+HIIT) (Active Comparator): Participants who do not receive nutritional education but are enrolled in a high-intensity interval training exercise program.
  Interventions: Other: The High-Intensity Interval Training (HIIT)
- Nutritional Education (EDU+INACT) (Active Comparator): Participants who receive nutritional education but not an exercise program.
  Interventions: Other: Behavioral: Nutritional education program
- Nutritional Education Moderate-intensity continuous training (EDU+MICT) (Experimental): Participants who receive nutritional education and are enrolled in a moderate-intensity continuous training exercise program.
  Interventions: Other: The Moderate-Intensity Continuous Training (MICT); Other: Behavioral: Nutritional education program
- Nutritional Education High-intensity interval training (EDU+HIIT) (Experimental): Participants who receive nutritional education and are enrolled in a high-intensity interval training exercise program.
  Interventions: Other: The High-Intensity Interval Training (HIIT); Other: Behavioral: Nutritional education program

INTERVENTIONS:
Other: The Moderate-Intensity Continuous Training (MICT) — 3 sessions per week in a cycle ergometer, with 1-2 days off between sessions, during a total of 12 weeks under the supervision of a personal trainer. MICT program will consist of sessions of approximately ˜45 min of moderate aerobic exercise (at the intensity at which the maximal fat oxidation was achieved in the laboratory test) in cycle ergometer.
  Arms: Moderate-intensity continuous training (CG+MICT); Nutritional Education Moderate-intensity continuous training (EDU+MICT)
Other: The High-Intensity Interval Training (HIIT) — 3 sessions per week in a cycle ergometer, with 1-2 days off between sessions, during a total of 12 weeks under the supervision of a personal trainer. HIIT program will consist of 3-5 series of 1 min duration at 90-130% of its maximum power (determined in the first training session), with 90 seconds of rest between sets (estimated total time of the session: 10 minutes). Depending on the number of training session, the load and the series will increase up to 40% more than the maximum load.
  Arms: High-intensity interval training (CG+HIIT); Nutritional Education High-intensity interval training (EDU+HIIT)
Other: Behavioral: Nutritional education program — The education intervention will consist of individual nutritional counselling. The nutritional education program will be conducted every 2 weeks for 12 consecutive weeks, with 20-min counselling sessions by an experienced nutritionist. Participants will be provided with an introduction (in an easy-to-understand manner) regarding the association between T2DM, gut microbiome and dietary habits. Firstly, the diet of the patient should be analysed, to determine which aspects can be improved, such as, total calories intake, amount and types of carbohydrates (highlighting the relevance of fibre), etc. Moreover, some suggestions about the combination of foods and culinary technical in order to manage the glycaemic index of foods will be provided. Finally, those pattern of the Mediterranean diet and some qualitative aspects and aids (as the size of the plat or avoid having the food platter on the table) will be taught the patients.
  Arms: Nutritional Education (EDU+INACT); Nutritional Education High-intensity interval training (EDU+HIIT); Nutritional Education Moderate-intensity continuous training (EDU+MICT)

SUMMARY:
We hypothesize that the combination of a nutritional education intervention with a HIIT-based physical exercise program improve muscle metabolism through positive modifications of gut microbiota in people with T2DM, leading to better glycaemia/insulinaemia levels, reduction of body fat mass and improving quality of life.

The project is a randomized controlled clinical trial in 120 participants with T2DM and obesity, which aims to determine the efficacy of a nutritional education program and the role of physical exercise type on health related variables. The participants will be of both sexes with age between 40 and 55 years, belonging to the Province of Cádiz. The design has two 12-week interventions; the main factor has 2 levels: participants who receive the nutritional education (EDU) and controls (CG); the second factor has 3 levels: high-intensity interval training (HIIT), moderate intensity continuous training (MICT), and controls (INACT). Therefore, participants will be randomized into 6 groups (n=20), adjusted by gender (≈50% in each group): EDU+HIIT, EDU+MICT, EDU+INACT, CG+HIIT, CG+MICT, CG+INACT.

The outcome variables, which will be measured before and after the intervention, will include: dietary intake assessment, physical activity assessment, quality of life, faecal samples, blood samples, blood pressure, appetite assessment, muscle biopsy samples, body composition and fluids, basal metabolism, maximal fat oxidation test and cardiorespiratory fitness.

DETAILED DESCRIPTION:
Approximately 500 million people have Type 2 Diabetes Mellitus (T2DM) in 2018 and it is expected to increase between 20% and 50% over the next 10 years. T2DM is also called non-insulin-dependent or adult-onset, and it results from the body's ineffective use of insulin, being the result of excess body weight and physical inactivity. Diabetes is the 7 leading cause of death by increasing the risks of cardiovascular and other diseases, many of which (43%) occur prematurely and are largely preventable through adoption of policies to create supportive environments for healthy lifestyles.

Improving the implementation of health-related education programs is a key tool for behaviour change; however, not all education supports behavioural change. The terms education and knowledge are often thought of interchangeably. Nevertheless, while knowledge is defined as "facts, information, and skills acquired by a person through experience or education", education is a comprehensive term that can be defined as "the process of receiving or giving systematic instruction" or as "an enlightening experience". Therefore, interventions should attempt the education achievement in order to improve healthy lifestyles and reduce diabetes prevalence, complications and morbimortality. In this line, the impact of nutritional counselling on weight reduction, glycaemia control, and improve of health in obese and diabetes population have been previously study with inconsistent results. Thus, education strategies should be optimized to achieve behaviour changes related to nutrition and physical exercise.

Recently it has been discover than gut microbiota can modulate behaviour, including nutritional behaviour and decisions, therefore, gut microbiota can have an impact on the efficacy of an education program. Gut microbiota is composed of more than 100 billion microorganisms classified in at least 1000 different species of bacteria, fungi, viruses and yeasts. In light of these considerations, Nobel laureate Joshua Lederberg proposed to consider the microbiota, especially the intestinal one, as a "superorganism". One of the great findings in neuroscience is the connection of the intestinal microbiota and the brain, called gut-brain axis, telling us whether to eat or not, even what food (for example the desire to eat something sweet or salty). These results can be a great advance for the area of education and behavioural sciences, especially of those education program focused on improve nutritional habits.

Moreover, even maintaining similar energy intake through diet and similar physical activity levels, a healthy change of gut microbiota is able to reduce body fat percentage, what has a positive impact on the prevention and treatment of T2DM. Therefore, educational programs focused on improving gut microbiota can be a useful tool to respond to the Global Plan of Action on Non-communicable Diseases, and could reduce the failure of some weight loss educational strategies and programs. Recently it has been shown that gut microbiota plays a significant role in the pathophysiology of T2DM modulating the secretion of insulin and glucose. Therefore, tools that establish the microbiota should be promoted, such as nutritional restoration strategies, through prebiotics and probiotics, in obesity and T2DM populations as we have previously study.

In addition, physical exercise seems to improve gut microbiota composition, specifically the Firmicutes spp. / Bacteroidetes spp. ratio, additionally, a positive correlation has been found between Lactobacillus spp. and Bifidobacterium spp. with serum leptin levels in trained rats. Most exercise programs to combat obesity have been based primarily on aerobic exercises. Aerobic training is associated with a decrease in body fat mass, especially visceral fat mass, increases insulin sensitivity, lowers baseline glucose and insulin levels, and increases the expression of glucose and fatty acid transport proteins in muscle fibres. Workouts that are performed at the intensity at which the person burns more fat (FatMax) seems to reduce body fat and insulin resistance in older women with type 2 diabetes. However, the time taken for these training sessions is approximately 60-90 minutes a day.

According to previous scientific research, we hypothesize that the combination of a nutritional education intervention with a HIIT-based physical exercise program improve muscle metabolism through positive modifications of gut microbiota in people with T2DM, leading to better glycaemia/insulinaemia levels, reduction of body fat mass and improving quality of life.

The project is a randomized controlled clinical trial in 120 participants with T2DM and obesity, which aims to determine the efficacy of a nutritional education program and the role of physical exercise type on health related variables. The participants will be of both sexes with age between 40 and 55 years, belonging to the Province of Cádiz. The design has two 12-week interventions; the main factor has 2 levels: participants who receive the nutritional education (EDU) and controls (CG); the second factor has 3 levels: high-intensity interval training (HIIT), moderate intensity continuous training (MICT), and controls (INACT). Therefore, participants will be randomized into 6 groups (n=20), adjusted by gender (≈50% in each group): EDU+HIIT, EDU+MICT, EDU+INACT, CG+HIIT, CG+MICT, CG+INACT.

The outcome variables, which will be measured before and after the intervention, will include: dietary intake assessment, physical activity assessment, quality of life, faecal samples, blood samples, blood pressure, appetite assessment, muscle biopsy samples, body composition and fluids, basal metabolism, maximal fat oxidation test and cardiorespiratory fitness.

ELIGIBILITY:
Inclusion Criteria:

* Non smoking
* Non-alcoholic (<3 standard drinks per day)
* Body mass index >25 kg/m maintaining the habitual dietary patterns without a body mass reduction higher than 2% during the last 6 months
* Not being insulin dependent
* Absence of injury, disease or disability or other known medical condition which could affect the ability to successfully participate in physical exercise tests
* Absence of cardiovascular disease (angina, peripheral or cerebro-vascular disease, etc.).
* Absence of neurologic and psychiatric diseases.
* Absence of respiratory diseases (pulmonary hypertension, Chronic obstructive pulmonary disease, etc.).
* Absence of other metabolic diseases (hyper/hypo parathyroidism, hyper/hypothyroidism, Cushing's disease, Type 1 diabetes, etc.)
* Absence of active inflammatory bowel disease
* Absence of kidney disease
* Absence of tumours
* Absence of coagulation dysfunction
* Not under treatment with medications k known to affect glucose metabolism, recent steroid treatment (within 6 months), or hormone replacement therapy
* Be able to understand a communication in Spanish or English.

Exclusion Criteria:

* They do not attend more than 2 or 4 consecutive sessions of nutritional counselling or physical training respectively.
* The lose more than 4 or 6 sessions in total of nutritional counselling or physical training respectively.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Assessed gut microbiota population | 12 weeks
  For the DNA extraction, fecal samples will be homogenized in a Stomacher-400 mixer. The DNA will be extracted using a mini QIAamp DNA stool kit (QIAGEN, Barcelona, Spain) as indicated by the manufacturer. Quantification is performed with a NanoDrop ND-1000 spectrophotometer (Thermo Fisher Scientific, DE, USA). For sequencing analysis, DNA extracted is amplified by Polymerase Chain Reaction (PCR). All PCRs will be performed in 25 μl of reaction volumes containing 12.5 μl of the KAPA HiFi Hotstart 2X prepared mixture (KAPA Biosystems, Woburn, MA), 5 μl of each direct and reverse primer (1 μM) and 2.5 μl of extracted DNA (10 ng) under standardized cycling conditions. PCR cleaning will be performed with beads and PCR products combined with AMPure XP beads (Beckman Coulter, USA). Determine gut microbiota composition and characterization, for classification of phylum, genus, and species of bacteria. Specifically the Firmicutes/Bacteroidetes ratio.
Assessed changes in Insulin Resistance | 12 weeks
  They will be determined using the ELISA technique for the concentration of insulin. The Homeostatic Model Assessment for Insulin Resistance insulin sensitivity index (HOMA-IR) will be calculated.
Muscle biopsy samples: mRNA expression by quantitative real-time PCR (Transcriptomic) | 12 weeks
  The mRNA levels of Glucose Transporter GLUT4, IRS1, PI 3-Kinase, PGC1-alpha, SIRT1, Mitofusin 1, Mitofusin 2, Complex I, III, IV, V of mitochondria (Nd1, Cyb, Co1, Atp6), CPT1B, and OPA1 will be analysed, for that, total RNA will be isolated from tissues (frozen muscle biopsies) an Illustra MiniRNA Spin kit (GE Healthcare). Then, cDNA will be obtained using a PrimeScript™ RT Master Mix (Perfect Real Time) (Takara), following the manufacturer's instructions. Relative quantification of mRNA will be performed using a Corbett RotorGene by using 6.5 ng of cDNA, forward and reverse primers at 100 nM each, and a SYBR Green PCR Master Mix Reagent kit (Life Technologies) in 10 μL of reaction. The mRNA levels will be normalized to those of housekeeping genes (b-actin, a-tubulin) and expressed as fold change.
Muscle biopsy samples: Western blot analysis (Proteomic) | 12 weeks
  Frozen muscle tissue will be homogenized in protein extraction buffer (RIPA buffer with phosphatase inhibitors and protease inhibitors). Protein concentration will be determined using a BCA protein assay kit (Thermoscientific). Then, samples will be separated on SDS-PAGE gels, and then transferred onto PVDF membranes (Millipore). The following primary antibodies will be used Rabbit polyclonal to PGC1 alpha, Rabbit monoclonal [EPR19274] to DRP1, Rabbit monoclonal [E104] to SIRT1, Rabbit monoclonal [EP2109Y] to AKT1 (phospho S473), Rabbit polyclonal to TIM44, Rabbit polyclonal to Glucose Transporter GLUT4, Rabbit polyclonal to IRS1, Rabbit polyclonal to AKT1, Rabbit monoclonal [EPR5683] to AMPK alpha 2 (phospho T172), Rabbit polyclonal to CPT1B, Total OXPHOS Human WB Antibody Cocktail, Rabbit polyclonal to Mitofusin 1, Rabbit polyclonal to OPA1, Mouse monoclonal [12C4F12] to MTCO2, Rabbit polyclonal to IRS1 (phospho S312), Rabbit polyclonal to AMPK alpha 2, Mouse monoclonal [6A
Muscle biopsy samples: Citrate synthase (CS) activity assay (Mitochondrial content marker) | 12 weeks
  Therefore, skeletal muscle (5 mg) will be homogenized in 100 μl cold CelLytic MT (Sigma) at pH 7.4 and protease inhibitor cocktail. The homogenized sample will be centrifuged at 12,000xg for 10 min and the supernatant containing the protein collected. After, 8 μg of protein, as determined by BCA protein assay. In addition to protein, the reaction mixture contained 1X assay buffer, 300 μM acetyl CoA and 100 μM 5,5'-Dithiobis-(2-nitrobenzoic acid). The reaction starts by adding 500 μM Oxaloacetate. CS activity is measured by continuous spectrophotometric rate determination at 412 nm, according to manufacturer instructions. Each sample will be run in triplicate.
Assessed changes from Appetite assessment | 12 weeks
  Since appetite feeling modulates nutritional behavior, the evaluation of appetite among the intervention groups can improve the quality of the study from a comprehensive perspective. After a period of 8-10 hours of fasting, an analog visual scale (AVS) will be completed in order to ensure the appetite felt by the participant in the morning. The AVS runs from 1 to 10, being the lowest value no appetite at all, and the maximum full appetite.
Assessed changes from Body composition: Fatmass and Fat-free mass. | 12 weeks
  Body composition will be estimated using a multifrequency bioimpedance of 8 electrodes previously validated (TANITAMC780MA). The calculation of impedance can estimate the fat mass and fat-free mass in kilograms. The patients will wear light clothing and will assume a posture in accordance with the manufacturers' instructions. Other previous considerations will be followed 24 hours before the measure: (i) to refrain from vigorous exercise, (ii) to take alcoholic drinks, (iii) to take energy drinks, and (iv) to be in a fasting state for at least 8 hours. Hydration status will be controlled through a urine color scale from clear to dark during the 7 days before assessment for adjusting variables.

SECONDARY OUTCOMES:
Assessed changes from dietary intake: Frequency of consumption | 12 weeks
  Dietary intake assessment by trained surveyors in a personal interview, using a Food Frequency Questionnaire (FFQ). The FFQ has been previously validated in Mediterranean population of Spain, and provides qualitative frequency of consumption over the last year. In addition, a semi-quantitative analysis of total energy, macro and micro nutrients will be performed. The results will be analysed through the DIAL® software for Windows, version 3.7.1.0, estimating the average of total energy in kilocalories, macro and micro nutrients in grams for each participant.
Assessed changes from dietary intakes: 24 hours dietary recalls | 12 weeks
  Dietary intake assessment by trained surveyors in a personal interview, using three 24h dietary recalls (24HR). The results will be analysed through the DIAL® software for Windows, version 3.7.1.0, estimating the average of total energy in kcal, macro and micro nutrients in grams for each participant.
Assessed changes from accelerometry: Physical activity time | 12 weeks
  Physical activity assessment will be carried out through accelerometers (direct method) at the wrist during 7consecutive days. The data generated by the accelerometers will be analysed by using ActiLife 6.6.2 software (ActiGraph, Florida; USA), using Freedson (1998) cut-points for adults and Choi's validation. The software calculates in the base the movements of the accelerometer's time of light, moderate, and vigorous physical activity in minutes.
Assessed changes from physical activity | 12 weeks
  Physical activity assessment will be estimated by the participant's self-reported International Physical Activity Questionnaire Short Version (IPAQ-SF) previously validated in Spain. The IPAQ-SF calculates moderate and vigorous activity time in minutes per week.
Assessed changes from resting fat oxidation | 12 weeks
  Basal Metabolism will be assessed to determine the Resting Fat Oxidation of each participant before and after the 12-week intervention, since its importance as a health indicator and relationship with obesity. Therefore, Oxygen uptake (VO2), carbon dioxide production (VCO2) will be registered at resting conditions on a bed in a supine position during 30 min. Resting indirect calorimetry will be measured using a gas analyser of an open circuit, Jaeger MasterScreen CPX® (CareFusion, San Diego, USA). Heart Rate will be measured continuously over the test with Polar Team 2 (Polar Electro Inc., Lake Success, NY). Resting Fat Oxidation in grams per minute will be calculated by the indirect equation proposed by Frayn.
Assessed changes from cardiorespiratory fitness | 12 weeks
  Maximum VO2 test: To determine the maximal oxygen consumption (VO2max) during exercise in liters per minute, a gradual test on cycloergometer (Lode Excalibur, Netherlands) will be performed. The gas exchange will be measured by Jaeger MasterScreen CPX® (CareFusion, San Diego, USA)The test will be continuing the MFO from the load when the respiratory quotient reaches a stable value of 1 or higher. Once this point is reached, 15 Watts increments will occur every minute until exhaustion is reached, until achieving the VO2max. Throughout the test a cadence of 80 r.p.m. will be maintained. Heart rate will be recorded in beats per minute.
Assessed changes from maximal fat oxidation | 12 weeks
  Maximal fat oxidation test (MFO) to determine the maximal fat oxidation during exercise (MFO), a gradual test on cycloergometer (Lode Excalibur, Netherlands) will be performed. The test will begin with a load of 15 Watts, increasing 15Watts every 3 minutes until the respiratory quotient reaches a stable value of 1 or higher. Throughout the test a cadence of 80 r.p.m. will be maintained. Calculation in the base of expired gases will be made for the estimation of grams per minute of fat oxidation.
Assessed changes from self-reported quality of life | 12 weeks
  Self-reported quality of life will be registered by applying the Short Form 36-health survey (SF-36) questionnaire previously validated in Spain. The SF-36 is a generic measure of quality of life and has been evaluated for a wide variety of medical conditions, including diabetes. The SF-36 includes 36 questions that evaluate 8 subscales, scores for each scale range from 0 to 100, with higher scores indicating higher level of function or wellbeing. The physical component summary is derived from the 4 subscales of physical functioning, role physical, bodily pain, and general health; while the mental component summary is derived from the subscales of vitality, social functioning, role emotional, and mental health.
Assessed changes from blood pressure | 12 weeks
  Systolic and diastolic blood pressures will be recorded three times by using the validated Omron HEM 742 blood pressure monitoring device with the participant seated, back supported in chair and feet flat on floor without legs crossed, after they rested 5 minutes. The guidelines of the Hypertension and Cardiology European Societies and the Spanish one will be used to classify blood pressure stages of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Gustavo Ponce González, PhD, Principal Investigator — University of Cádiz; Cristina Casals, PhD, Principal Investigator — University of Cádiz
Locations (1):
- Facultad de Ciencias de la Educación, Puerto Real, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No